CLINICAL TRIAL: NCT04881292
Title: Reference Values of Carotid Intima-media Thickness and Arterial Stiffness in Chinese Adults Based on Ultrasound Radio Frequency Signal: A Nationwide, Multicenter Study
Brief Title: RF Based QIMT & QAS Study on Chinese Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Esaote (Shenzhen) Medical Equipment Co. Ltd (Unknown); Zhejiang University (Other); Shannxi Provincial People's Hospital (Unknown); Shengjing Hospital (Other); First Hospital of China Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Beijing University of Chinese Medicine Third Affiliated Hospital (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology (Unknown); The First Hospital of Jilin University (Other); The Afffiliated Hospital of Guizhou Medical University (Unknown); Yan An Hospital Affiliated to Kunming Medical University (Unknown); Second Affiliated Hospital of Guangzhou Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Ruijin Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Anhui Medical University (Other); The First Affiliated Hospital of USTC (Unknown); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Hospital of Northwestern Polytechnical University (Unknown); GEM Flower Xian Changqing Staff Hospital (Unknown); Xi'an Central Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Karamay Central Hospital of Xinjiang (Unknown); Fourth Affiliated Hospital of Xinjiang Medical University (Other); Xi'an No.1 Hospital (Unknown); Xianyang Hospital of Yan'an University (Unknown); General Hospital of Xinjiang Production and Construction Corps (Unknown); Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Lijun Yuan, MD, PhD, Director of the department of ultrasound diagnostics, Tang-Du Hospital
Other Study IDs: 20210402V2.0
Record Dates: First submitted 2021-05-01; First posted 2021-05-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Healthy; Adults; Carotid Intima-media Thickness; Vascular Stiffness; Chinese

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to establish the normal reference values of carotid artery intima-media thickness and vascular elasticity of Chinese adults based on ultrasound radio frequency technology through a multi-center large-sample study, which provides important information for the risk prediction and prognosis evaluation of Chinese adults' cardiovascular disease.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will undergo a one-time examination of vascular ultrasound, including general characteristics and the target ultrasound parameters.

To detect the smallest difference between adjacent age groups within the age range 18-79 (6 groups, α = 0.05, β = 0.20, Statistical Power = 0.80). Given the influence of multiple centers, the minimum sample size is 1800, the optimal sample size is 3500. The male to female ratio is 1:1.

Quality Control including the pre-study training and data monitoring during the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-79
* The blood pressure is normal: systolic blood pressure <140 mmHg, and diastolic blood pressure <90 mmHg
* The physical examination and electrocardiogram are normal

Exclusion Criteria:

* Subjects with carotid intima-media thickness ≥ 1.0 mm should be excluded;
* Subjects with previous cardiovascular disease history and medication history should be excluded. The main diseases include coronary heart disease, congenital heart disease, heart failure, hypertension, stroke, hyperlipidemia, diabetes, aortic arteritis, etc.;
* Subjects with past medical history and medication history of endocrine, rheumatism, chronic respiratory disease, liver and kidney disease should be excluded;
* Obese subjects (BMI ≥ 28 kg/m2), professional athletes, pregnant and lactating women should be excluded;
* Alcohol or drug addicts and smokers who have not quit smoking should be excluded.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Han Chinese adults
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Intima-media thickness | one-time measurement on the day of ultrasound examination
  millimeter, one-time measurement throughout the study
Carotid stiffness index | one-time measurement on the day of ultrasound examination
  =D▪ln(Ps/Pd)/ΔD, D: diastolic carotid diameter; Ps, systolic pressure; Pd, diastolic pressure; ΔD: Change of diameter in systolic. one-time measurement throughout the study
Pulse wave velocity | one-time measurement on the day of ultrasound examination
  m/sec,one-time measurement throughout the study
Artery compliance coefficient | one-time measurement on the day of ultrasound examination
  mm2kPa-1; =π▪(2▪D▪ΔD+ΔD2)/4▪ΔP; D: Diastolic diameter; ΔD: Change of diameter in systolic; ΔP, pulse pressure. one-time measurement throughout the study
Age | one-time measurement on the day of ultrasound examination
  years, one-time measurement throughout the study

SECONDARY OUTCOMES:
blood pressure | one-time measurement on the day of ultrasound examination
  mmHg, one-time measurement throughout the study
fasting blood glucose | one-time measurement with 7 days before or after ultrasound examination
  mmol/L, one-time measurement throughout the study
Total cholesterol | one-time measurement with 7 days before or after ultrasound examination
  mmol/L, one-time measurement throughout the study
Triglycerides | one-time measurement with 7 days before or after ultrasound examination
  mmol/L, one-time measurement throughout the study
Height | one-time measurement on the day of ultrasound examination
  m, one-time measurement throughout the study
Weight | one-time measurement on the day of ultrasound examination
  kg, one-time measurement throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Yuan, PhD; MD, Principal Investigator — Tangdu Hospital-Air Force Medical University
Locations (34):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Air Force Medical Center, Beijing, Beijing Municipality
  - Beijing University of Chinese Medicine Third Affiliated Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Afffiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Air Force Medical University, Xi'an, Shannxi
  - Shannxi Provincial People's Hospital, Xi'an, Shannxi
  - GEM Flower Xian Changqing Staff Hospital, Xi'an, Shannxi
  - Hospital of Northwestern Polytechnical University, Xi'an, Shannxi
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi
  - The Second Affiliated Hospital of Xi'an Medical University, Xi'an, Shannxi
  - Xi'an Central Hospital, Xi'an, Shannxi
  - Xi'an No.1 Hospital, Xi'an, Shannxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - General Hospital of Xinjiang Production and Construction Corps, Ürümqi, Xijiang
  - Karamay Central Hospital of Xinjiang, Karamay, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Fourth Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yan An Hospital Affiliated to Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place